CLINICAL TRIAL: NCT03056677
Title: Does Modified Whey Protein Lower Post Meal Glucose Levels
Brief Title: Modified Whey Protein and Effect on Post Meal Glucose Levels Study
Acronym: MWPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aberdeen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 2016/RINH/1
Record Dates: First submitted 2017-02-07; First posted 2017-02-17 (Actual); Last update posted 2018-12-12 (Actual); Status verified 2018-12

CONDITIONS: Metabolism Disorder, Glucose
Keywords: Whey protein; Dietary supplementation; Glucose; GLP-1; Satiety
MeSH Terms: conditions — Glucose Metabolism Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Experimental): No Whey Protein
  Interventions: Dietary Supplement: Control
- Normal Whey protein (Experimental): Whey protein (50grams) drink will be given prior to a mixed carbohydrate meal
  Interventions: Dietary Supplement: Normal Whey protein
- Modified Whey (Experimental): Modified whey protein will be given
  Interventions: Dietary Supplement: Modified whey protein

INTERVENTIONS:
Dietary Supplement: Control — 200mls water will be given prior to a mixed carbohydrate meal
  Arms: Control
Dietary Supplement: Normal Whey protein — Whey protein (50grams) drink will be given prior to a mixed carbohydrate meal
  Arms: Normal Whey protein
Dietary Supplement: Modified whey protein — Modified whey protein (50grams) drink will be given prior to a mixed carbohydrate meal
  Arms: Modified Whey

SUMMARY:
After meals, the level of glucose rises in the circulation. In some individuals who are overweight and older, blood glucose can rise to levels which can damage tissues and cause health problems. Usually the hormone insulin, released from the pancreas, effectively lowers blood glucose. However, in overweight and older people insulin is less effective. Certain foods can lower the rise in blood glucose, particularly proteins. This works by increasing the release of a hormone from the gut called Glucagon-Like Peptide 1 (GLP-1), which in turn increases the release of insulin. A Component of milk left over after cheese making, termed Whey protein, is particularly good at releasing GLP-1. Whey protein is used as a food additive and taken as a supplement to help build muscle. Whey protein is a mixture of proteins which the investigators have modified to be more effective at lowering blood glucose. Using laboratory tests the investigators identified a protein present in Whey that does not increase levels of GLP-1 and removed it. It's removal raises the levels of other proteins which are more effective. In this study, the investigators would like to test the effectiveness of the "modified" whey protein. To do this, 30 older, overweight volunteers will be recruited and given the modified whey protein, a normal whey protein or a mixture of amino acids and then a breakfast meal to raise their blood glucose levels. These drinks will be given in a randomised sequence 1 week apart. On each visit, blood samples to measure blood glucose and related hormone levels will be taken. As GLP-1 can also have an effect on appetite, the investigators will measure the effect of the modified whey protein on subsequent appetite in the volunteers by asking them how hungry they feel.

DETAILED DESCRIPTION:
The prevalence of obesity and associated type 2 diabetes has risen dramatically, adversely affecting health and life expectancy and increasing health care costs. There is an urgent need to lower the incidence or delay the onset of both conditions by lifestyle-related interventions. Dietary whey protein acts in the gut to release GLP-1 and insulin release, thereby lowering post-meal glucose levels and satiety. Whey protein is a mixture of proteins which the investigators have modified to be potentially more effective at lowering blood glucose. Using laboratory tests, a protein present in whey that does not increase levels of GLP-1 was identified and removed. Its removal raises the levels of other proteins which are more effective. The study will test the effectiveness of the "modified" whey protein. If the modified whey protein is found to be more effective it may be used to minimise the post-meal rise in glucose levels.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women aged 55-75years
* Body Mass index range from 25-35 kg/m2
* Blood pressure below 160/90mmHg

Exclusion Criteria:

* Milk or milk protein allergy
* Lactose Intolerance
* Diabetes
* Smoking
* Taking anoretic drugs, steroid medications, medications known to affect gastric motility or any hypoglycaemic agents
* Unsuitable veins for venous blood sampling
* Inability to spell, read and understand the English language

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-08 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Insulin response | 18months
  Post supplementation levels of glucose will be measured to assess insulin response

SECONDARY OUTCOMES:
Insulin Concentration | 18 months
  Post supplementation levels of Insulin will be measured to assess insulin response
GLP-1 level | 18months
  Post supplementation levels of GLP-1 will be measured to assess insulin response
C-peptide levels | 18months
  Post supplementation levels of C-peptide will be measured to assess insulin response
Increased satiety using a visual analogue scale | 5 hours
  At baseline and 3 hours post consumption satiety will be measured by completion of a visual analogue scale questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Lynda Williams, BSc, PhD, Principal Investigator — University of Aberdeen
Locations (1):
- University of Aberdeen, The Rowett Institute, Aberdeen, United Kingdom

IPD SHARING:
Plan to Share IPD: No